CLINICAL TRIAL: NCT04759573
Title: Effects of Early Vocal Contact (EVC) in the Neonatal Intensive Care Unit: A Multi-centre, Randomized Clinical Trial
Brief Title: Effects of Early Vocal Contact (EVC) in the Neonatal Intensive Care Unit
Acronym: EVC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Elisa Della Casa Muttini (Other)
Responsible Party: Sponsor-Investigator, Elisa Della Casa Muttini, Principal Investigator, Azienda Ospedaliero-Universitaria di Modena
Organization: Azienda Ospedaliero-Universitaria di Modena (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Early Vocal Contact
Record Dates: First submitted 2021-02-06; First posted 2021-02-18 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Early Intervention; Prematurity
Keywords: Early Vocal Contact; Neonatal Intensive Care Unite; Preterm Infants
MeSH Terms: conditions — Premature Birth | interventions — Behavior Observation Techniques

STUDY DESIGN:
Intervention Model Description: A four-site randomized controlled trial will be conducted to investigate the short- and long-term physiological and neurobehavioral effects of Early Vocal Contact.
Who Masked: Outcomes Assessor
Masking Description: The intervention is performed by mothers who have to administer the speech or singing or they have to observe.
  The research assistant will support mothers to deliver the intervention The outcome assessors will be blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Vocal Contact (Experimental): The EVC will take place in the hospital room while infants are in their individual incubators or open cribs. In the intervention group, mothers will be asked to speak and sing to their infants continuously over a 10-min period for each type of intervention (20 min in total). Mothers will be asked to talk in their native language and to sing familiar songs, while observing their infant's reactions. The order of the two vocalizations, speaking and singing, will be reversed in the next intervention.
  Early Vocal Contact will be performed by mothers three times a week for 2 weeks, more than one hour after afternoon feeding. It will begin when the newborns are in an active sleep state, in calm awake state or in active awake state, but not in deep sleep or crying. Preterm infants will be enrolled from 25+0 to 32+6 weeks of GA, following the established inclusion criteria.
  Interventions: Behavioral: Early Vocal Contact
- Behavioral observation (Active Comparator): Mothers in the active control group will be encouraged to spend the same amount of time next to the incubator, observing the infant's behaviours through a standard cluster of indicators.
  Interventions: Behavioral: Behavioral Observation

INTERVENTIONS:
Behavioral: Early Vocal Contact — Mothers will be asked to speak and sing to their infants continuously over a 10-min period for each type of intervention (20 min in total). Mothers will be asked to talk in their native language and to sing familiar songs, while observing their infant's reactions. The order of the two vocalizations, speaking and singing, will be reversed in the next intervention.
  Arms: Early Vocal Contact
Behavioral: Behavioral Observation — Mothers in the active control group will be encouraged to spend the same amount of time next to the incubator, observing the infant's behaviours through a standard cluster of indicators.
  Arms: Behavioral observation

SUMMARY:
Background: Preterm infants are at risk for developing altered trajectories of cognitive, social, and linguistic competences compared to a term population. This is mainly due to medical and environmental factors, as they are exposed to an atypical auditory environment and, simultaneously, to long periods of early separation from their parents. The short-term effects of Early Vocal Contact (EVC) on an infant's early stability have been investigated, but currently, there is limited evidence of its impact on the infant's autonomic nervous system maturation, as indexed by the heart rate variability, as well as on its long-term impact on infant neurodevelopment. This multi-centric study aims to investigate the effects of EVC on a preterm infant's physiology, neurobehaviour, and development.

Methods: Eighty stable preterm infants, born at 25 to 32 weeks and 6 days gestational age, without specific abnormalities, will be selected and randomized to either an intervention or a control group. The intervention group will receive EVC: mothers talking and singing to their preterm infants for 10 minutes thrice a week for 2 weeks. Mothers in the control group will be encouraged to spend the same amount of time next to the incubator, observing the infant's behaviour through a standard cluster of indicators. Infants will be assessed at baseline, at the end of the intervention, at term equivalent age, and at 3, 6, 12- and 24-months corrected age, with a battery of physiological, neurobehavioral, and developmental measures.

Discussion: Early interventions in the neonatal intensive care unit have shown important effects on the neurodevelopment of preterm infants, lowering the negative long-term effects of an atypical auditory and interactional environment. This study will provide new insights into the mother-infant early contact as protective intervention against the sequelae of prematurity during the sensitive period of development. An early intervention, such as EVC, is intuitive and easy to implement in the daily care of preterm infants. However, its long-term effects on infant neurodevelopment and on maternal sensitivity and stress still need accurate investigations.

DETAILED DESCRIPTION:
Aims This study aims to test the effects of EVC on infants born prematurely between 25 and 32 weeks and 6 days GA.

The effects on newborns will be assessed at physiological (primary outcome), neurobehavioral, and developmental levels during the intervention, at term equivalent age, and at 12- and 24-months CA. The effect of EVC will also be assessed on maternal stress at hospital discharge and on the mother's presence in the NICU.

Design A four-site randomized controlled trial will be conducted to investigate the short- and long-term physiological and neurobehavioral effects of EVC.

Participants Eighty preterm infants, born at 25 to 32 weeks and 6 days GA, will be recruited from the four centres (20 per centre).

Recruitment will be undertaken in each centre by a trained research assistant (RA), who will review birth records daily. After obtaining permission from the attending physicians of both the mother and the infant, the RA will invite qualifying families to participate in the study and will obtain written informed consent from those enrolling. Infants will be then assigned to the EVC intervention or control group using a randomized design, stratifying infants by gender and GA (see Randomization). Mothers whose infants are assigned to the control group will be asked to spend the same amount of time as that of mothers in the intervention group, observing their infants' spontaneous behaviour, with the subsequent compilation of an observation grid developed ad hoc, according to few indicators drawn from The Neonatal Behavioural Assessment Scale (NBAS).

ELIGIBILITY:
Inclusion Criteria:

* • GA between 25+0 and 32 +6 weeks at birth

  * Apgar score: ≥ 7 at 10 minutes
  * Birth weight: >3th centile and <97th centile
  * Birth cranial circumference: >10th centile
  * Periventricular leukomalacia (PVL) grade 1
  * Intraventricular haemorrhage (IVH) grade 1-2
  * Hypoglycaemia
  * Hyponatremia acceptable, provided they are not persistent and severe
  * Hypocalcaemia

Exclusion Criteria:

* • PVL, grade III and IV

  * IVH, grade III and IV
  * Sepsis (vertical and horizontal)
  * Congenital malformations and/or genetic abnormalities
  * Need of respiratory support with high flow/nCPAP
  * Repeated apnoea associated with bradycardia and fall of saturation
  * Hyaline membrane disease
  * Respiratory Distress Syndrome
  * Hyperbilirubinemia, requiring exchange transfusions during hospitalization
  * Lack of informed consent signed by the parents

The exclusion criteria for the mothers will be:

* Presence of depressive symptoms
* Drug abuse
* Age ˂18 years

Ages: 25 Weeks to 33 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in Heart Rate Variability | Pre intervention (baseline), during the intervention and immediately after the intervention
  Heart rate is the number of heartbeats per minute.

SECONDARY OUTCOMES:
Change in General Movement Assessment | Pre intervention (baseline)
  The General Movement quality from video recording will be scored according to the Ferrari optimality score. Two blinded coders will attribute a single final score for each infant at each time point. For each item a description of optimal performance is given and scored with "2" (e.g., cramped components are absent). Less optimal performance is scored with "1" (e.g., cramped components are occasionally present); non-optimal performance is scored with "0" (e.g., cramped components are predominately present).
  Adding the scores of each item within a category ("neck and trunk", "upper extremity" and "lower extremity") plus the score for "sequence" gives the GM optimality score with a minimum value of 5 and a maximum value of 42, indicating optimal performance. The minimum score (worst performance) is 5.
Change in General Movement Assessment | After the intervention, at Term Equivalent Age
  The General Movement quality from video recording will be scored according to the Ferrari optimality score. Two blinded coders will attribute a single final score for each infant at each time point. For each item a description of optimal performance is given and scored with "2" (e.g., cramped components are absent). Less optimal performance is scored with "1" (e.g., cramped components are occasionally present); non-optimal performance is scored with "0" (e.g., cramped components are predominately present).
  Adding the scores of each item within a category ("neck and trunk", "upper extremity" and "lower extremity") plus the score for "sequence" gives the GM optimality score with a minimum value of 5 and a maximum value of 42, indicating optimal performance. The minimum score (worst performance) is 5.
Change in General Movement Assessment | At 3 months
  The General Movement quality from video recording will be scored according to the Ferrari optimality score. Two blinded coders will attribute a single final score for each infant at each time point. For each item a description of optimal performance is given and scored with "2" (e.g., cramped components are absent). Less optimal performance is scored with "1" (e.g., cramped components are occasionally present); non-optimal performance is scored with "0" (e.g., cramped components are predominately present).
  Adding the scores of each item within a category ("neck and trunk", "upper extremity" and "lower extremity") plus the score for "sequence" gives the GM optimality score with a minimum value of 5 and a maximum value of 42, indicating optimal performance. The minimum score (worst performance) is 5.
The Griffiths Mental Development Scales (GMDS) | At 6 months corrected age
  The GMDS will be assessed with mean values in 4 subscales (Locomotor, Per-Social, Hear/Speech, Hand/Eye). A composite final Performance score will also be assessed for each participant at each time point. The mean values will be compared between the intervention and control groups. Scores range from 0 to 109, with better results with higher values.
The Griffiths Mental Development Scales (GMDS) | At 12 months corrected age
  The GMDS will be assessed with mean values in 4 subscales (Locomotor, Per-Social, Hear/Speech, Hand/Eye). A composite final Performance score will also be assessed for each participant at each time point. The mean values will be compared between the intervention and control groups. Scores range from 0 to 109, with better results with higher values.
MacArthur-Bates Communicative Development Inventories | At 12 months (Gestures and Words Form) and 24 months (Words and Sentences Form) corrected age.
  Each child, at each time point, will receive a final score for each questionnaire, measured as a discrete numeric value; the mean values will be compared in the intervention and control groups. The minimum score il 0 and the maximum is 429, with higher scores for better performance.
MacArthur-Bates Communicative Development Inventories | At 12 months corrected age
  Each child, at each time point, will receive a final score for each questionnaire, measured as a discrete numeric value; the mean values will be compared in the intervention and control groups. The minimum score il 0 and the maximum is 429, with higher scores for better performance.
MacArthur-Bates Communicative Development Inventories | At 24 months corrected age
  Each child, at each time point, will receive a final score for each questionnaire, measured as a discrete numeric value; the mean values will be compared in the intervention and control groups. The minimum score il 0 and the maximum is 429, with higher scores for better performance.
Parole in Gioco (PinG) test | At 24 months corrected age
  Linguistic test for assessing lexical comprehension and production for early childhood. The minimum score il 0 and the maximum is 60, with higher scores for better performance.
Change in Parental Stressor Scale (PSS-NICU) | Pre intervention
  The PSS-NICU aims at assessing the parental perception of stressors derived from the physical and psycho-social environment of the NICU across three domains: (i) their parental role, (ii) their infant's behaviour and appearance, and (iii) the sights and sounds in the NICU. For each domain, a mean score will be assessed, and a final composite stress score will be calculated from the mean values of the single scores. Each mother, at each time point, will receive a final score for the single questionnaire (range 0-10). The minimum score il 0 and the maximum is 156, with lower scores for better mental health levels.
Change in Parental Stressor Scale (PSS-NICU) | At hospital discharge
  The PSS-NICU aims at assessing the parental perception of stressors derived from the physical and psycho-social environment of the NICU across three domains: (i) their parental role, (ii) their infant's behaviour and appearance, and (iii) the sights and sounds in the NICU. For each domain, a mean score will be assessed, and a final composite stress score will be calculated from the mean values of the single scores. Each mother, at each time point, will receive a final score for the single questionnaire (range 0-10). The minimum score il 0 and the maximum is 156, with lower scores for better mental health levels.
Maternal presence in the NICU | At hospital discharge
  Time that the mothers spend in the NICU (hours) using maternal self-report forms will be filled out after each visit to the NICU

CONTACTS AND LOCATIONS:
Locations (1):
- Uiversity Hospital of Modena and Reggio Emilia, Modena, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Filippa M, Devouche E, Arioni C, Imberty M, Gratier M. Live maternal speech and singing have beneficial effects on hospitalized preterm infants. Acta Paediatr. 2013 Oct;102(10):1017-20. doi: 10.1111/apa.12356. Epub 2013 Aug 8. PMID 23848529
- [Result] Filippa M, Lordier L, De Almeida JS, Monaci MG, Adam-Darque A, Grandjean D, Kuhn P, Huppi PS. Early vocal contact and music in the NICU: new insights into preventive interventions. Pediatr Res. 2020 Jan;87(2):249-264. doi: 10.1038/s41390-019-0490-9. Epub 2019 Jul 2. PMID 31266053
- [Derived] Filippa M, Nardelli M, Sansavini A, Meloni S, Picciolini O, Lunardi C, Cecchi A, Corvaglia L, Grandjean D, Scilingo EP, Della Casa E, Berardi A; EVC Group; Ferrari F. Maternal singing sustains preterm hospitalized newborns' autonomic nervous system maturation: an RCT. Pediatr Res. 2024 Mar;95(4):1110-1116. doi: 10.1038/s41390-023-02932-4. Epub 2023 Dec 6. PMID 38057574
- [Derived] Filippa M, Della Casa E, D'amico R, Picciolini O, Lunardi C, Sansavini A, Ferrari F. Effects of Early Vocal Contact in the Neonatal Intensive Care Unit: Study Protocol for a Multi-Centre, Randomised Clinical Trial. Int J Environ Res Public Health. 2021 Apr 8;18(8):3915. doi: 10.3390/ijerph18083915. PMID 33917889